CLINICAL TRIAL: NCT03742661
Title: Impact of SPEAC® System Data on Therapeutic Decisions Related to Convulsive Seizure Patients With a New Diagnosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brain Sentinel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CPT-03-2018
Record Dates: First submitted 2018-08-02; First posted 2018-11-15 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Participating physicians will recruit patients meeting the inclusion and exclusion criteria. Upon completion of screening and enrollment procedures study participants will be randomly assigned to one of two groups using a randomized call-in system: treatment or standard of care.
  Demographics will be obtained for both groups during this initial clinic visit. The treatment group will be prescribed the Brain Sentinel® SPEAC System for use in the home environment. Study Participants in the standard of care group will be given standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): SPEAC System
  Interventions: Device: SPEAC System
- Standard of Care (No Intervention): Standard of Care

INTERVENTIONS:
Device: SPEAC System — Surface Electromyography (sEMG) based seizure monitoring and alerting system
  Other Names: Brain Sentinel Monitoring and Alerting System
  Arms: Treatment Group

SUMMARY:
This is an open label, randomized, prospective study of the impact on healthcare utilization of a surface Electromyography (sEMG) based seizure monitoring and alerting system for Veterans with a history of motor seizures (epileptic, non-epileptic or unknown) with upper extremity motor involvement, presenting with questionable spell characterization, taking place in the home setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a veteran with a reported history of motor seizures (epileptic, non-epileptic or unknown) with upper extremity motor involvement, presenting with questionable spell characterization.
2. Subjects has failed fewer than 3 anti-epileptic drugs (single or combination).
3. Male or Female between the ages 22 to 99.
4. If female and of childbearing potential, subject must agree to not become pregnant during the trial.
5. Can understand and sign written informed consent or will have a legally authorized representative (LAR) who can do so, prior to the performance of any study assessments.
6. Subject or Primary Caregiver must be competent to follow all study procedures.
7. Subject must be willing to use the Seizure Monitoring and Alerting System for a prolonged period of time (up to 120 days), for a minimum of 30 hours/ week.

Exclusion Criteria:

1. The subject cannot be pregnant, or nursing.
2. The subject cannot be sensitive or allergic to adhesives or tapes.
3. The subject may not be enrolled in another Clinical Trial.
4. The subject is homeless or in a home without a power supply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Impact Form Questionnaire | Up to 5 months
  The physician will complete this questionnaire after each 30 days of device use to determine if information acquired will change the physician's assessment of the patient's seizures and their treatment plan.

SECONDARY OUTCOMES:
Personal Impact of Epilepsy Scale (PIES) Survey | 1 year
  The PIES survey creates a composite score that can be used to assess the quality of life of patients with epilepsy, as well as sub-scales for assessing the quality of life in specific areas of life with epilepsy.
VR-12 Survey | 1 year
  This measure has been used in cost-effectiveness analyses and can be used to calculate quality adjusted life years (QALY).
Personal Impact of Epilepsy Scale (PIES) Survey | 5 years
  The PIES survey creates a composite score that can be used to assess the quality of life of patients with epilepsy, as well as sub-scales for assessing the quality of life in specific areas of life with epilepsy.
VR-12 Survey | 5 years
  This measure has been used in cost-effectiveness analyses and can be used to calculate quality adjusted life years (QALY).
VA Administrative Data | 1 year
  VA administrative data will be used to evaluate health outcomes.
VA Administrative Data | 5 years
  VA administrative data will be used to evaluate health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Bashir Shihabuddin, MD, Principal Investigator — Central Arkansas VA Medical Center
Locations (1):
- Lexington VA Medical Center, Lexington, Kentucky, United States